CLINICAL TRIAL: NCT02126605
Title: Accuracy of Blood Glucose Detection by Diabetes Alert Dogs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Linda Gonder-Frederick, Associate Professor, University of Virginia
Other Study IDs: 17296
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Type I Diabetes Mellitus
Keywords: diabetes alert dogs; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Even though there is growing interest in and use of trained Diabetes Alert Dogs (DADs) as a way to monitor blood glucose in type 1 diabetes (T1D), no scientific studies have confirmed the ability of DADs to accurately detect extreme high and low blood sugar. The current project is the first preliminary investigation into the accuracy of DADs, using scientifically rigorous research methods similar to those required to demonstrate accuracy in blood glucose meters. The primary aim of the project is to test the hypotheses that DADs are accurate at detecting extreme blood sugar levels in adults and children with T1D. The proposed project has several other secondary aims, which include determining: 1) the glycemic thresholds and time course for hypo- and hyperglycemic DAD alerts, 2) the degree to which alert accuracy is consistent across different DADs, and 3) whether or not DAD owners appear to experience better psychosocial status and quality of life compared to other individuals with T1D.

DETAILED DESCRIPTION:
In the proposed project, DAD alerts will be compared to blood glucose (BG) readings from a continuous glucose monitoring (CGM) device, as well as a BG meter. CGM, BG meter, and DAD alert data will be collected over a 4-wk period. CGM devices will be "blinded" so that BG readings will not be shown. This will allow for a direct comparison between objective glucose readings generated by approved BG monitoring devices and DAD alerts. This study will also utilize two methods for measuring DAD alerts: (1) use of the event recorder mechanism of the CGM device, and (2) collection of more detailed and qualitative data on DAD alerts using diaries (Daily DAD Diaries) to collect information concerning the occurrence, timing, and type of DAD alerts.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have had type 1 diabetes for at least 1 year and been taking insulin since diagnosis
* The participant must have a DAD placed in their home for a minimum of 6 months.
* Participants must not currently be using a continuous glucose monitor (CGM) in their diabetes management.
* Participants must be capable of performing all tasks involved in the study protocol, including filling out questionnaires and diaries in English.
* Participants must have an internet-connected computer compatible with study software.
* Willingness to avoid consumption of acetaminophen-containing products for the duration of the study.

Exclusion Criteria:

* Pregnant women-self reported
* Current use of a CGM
* History of a systemic deep tissue infection with methicillin-resistant staph aureus or Candida albicans

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetes Alert Dog (DAD) owners who have obtained their dogs from a specific training organization.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Percent agreement between DAD alerts and glucose readings | 5 weeks

SECONDARY OUTCOMES:
Psychosocial variables (quality of life, fear of hypo-/hyperglycemia, diabetes distress, self-efficacy, and DAD experiences) | Baseline, 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linda Gonder-Frederick, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Behavioral Medicine Research, Charlottesville, Virginia, United States